CLINICAL TRIAL: NCT06975618
Title: A Phase I/II, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Efficacy of CYH33 (a Selective PI3Kα Inhibitor) in Patients With PIK3CA-related Overgrowth Spectrum (PROS) and PIK3CA-related Vascular Malformations (PRVM)
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CYH33 in Patients With PIK3CA-related Overgrowth Spectrum (PROS) and PIK3CA-related Vascular Malformations (PRVM)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYH33-G208
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: PIK3CA-Related Overgrowth Spectrum (PROS); PIK3CA-related Vascular Malformations (PRVM)
MeSH Terms: interventions — CYH33

STUDY DESIGN:
Masking Description: The Phase I and Phase II PROS cohorts are both open-label, whereas the Phase II PRVM cohort is double-blind, with participants, care providers, investigators and outcome assessors unaware of the treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1：Adult cohort:； (Experimental): Phase I Adult Cohort: Adult patients with PIK3CA-related overgrowth spectrum (PROS) or PIK3CA-related vascular malformations (PRVM) will receive escalating oral doses of CYH33 to determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D). Expansion cohorts may be opened to further assess safety, tolerability, pharmacokinetics, and preliminary efficacy.
  Interventions: Drug: CYH33
- Arm 2: Phase I Adolescent Cohort (Experimental): Phase I Adolescent Cohort: Adolescent patients with PIK3CA-related overgrowth spectrum (PROS) or PIK3CA-related vascular malformations (PRVM) will receive escalating oral doses of CYH33 to determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D). Expansion cohorts may be opened to further assess safety, tolerability, pharmacokinetics, and preliminary efficacy.
  Interventions: Drug: CYH33
- Arm 3 : Phase II PROS Cohort (Experimental): Phase II PROS Cohort: An open-label, single-arm cohort. Adult and adolescent patients with PROS will receive CYH33 at RP2D. Dose escalation may be allowed based on tolerability and clinical assessment. Treatment will continue until disease progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: CYH33
- Arm 4 : Phase II PRVM Cohort (Experimental): Phase II PRVM Cohort: Adult and adolescent patients with PRVM will be randomized 2:1 to CYH33 or placebo during double-blind period. After 8 weeks of treatment, all patients will enter an open-label extension phase to receive CYH33. Treatment continues until disease progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: CYH33; Drug: Placebo

INTERVENTIONS:
Drug: CYH33 — CYH33: Participants will receive oral CYH33 once daily. The starting dose for adults in Phase I is 10 mg QD; adolescents begin at 5 mg QD. In Phase II, patients will receive RP2D determined in the Phase I study.
Drug: Placebo — Placebo: Matching placebo tablets will be administered once daily during the double-blind period of the Phase II PRVM cohort. Patients randomized to placebo will switch to CYH33 at the end of the blinded phase.
  Arms: Arm 4 : Phase II PRVM Cohort

SUMMARY:
This study is a multi-center, open-label, single arm, phase I/II study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of CYH33 in patients with PIK3CA-related overgrowth spectrum (PROS) and PIK3CA-related vascular malformations (PRVM)

ELIGIBILITY:
Key inclusion criteria:

1. The patient or the patient's legal guardian (if applicable) voluntarily signs the Informed Consent Form.
2. At the time of signing the informed consent, adult patients should be ≥18 years old (or meet the legal adult age according to local regulations), and adolescent patients should be ≥12 years old and <18 years old (or meet the legal definition of adolescent according to local regulations; additionally, adolescent patients should weigh ≥35 kg).
3. The patient is diagnosed with PIK3CA-related overgrowth spectrum (PROS) or PIK3CA-related vascular malformations (PRVM), and provides a report confirming PIK3CA mutation detected by local laboratory or the Sponsor-designated central laboratory, with at least one measurable lesion related to PROS or PRVM.
4. Patients should demonstrate adequate organ and bone marrow function during the 28-day screening period.

Key exclusion criteria:

1. PROS patients presenting solely with isolated macrodactyly, epidermal nevi/nevus, and megalencephaly (only one clinical feature or any combination of these three features) without other PROS-related lesions.
2. Patients who have received any systemic treatment for PROS or PRVM within 8 weeks prior to the first dose of study drug, or any drug treatment for PROS or PRVM (e.g., mTOR inhibitors) within 28 days prior to the first dose of study drug.
3. Patients who have previously received any PI3K inhibitor treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: The maximum tolerated dose (MTD) and/or phase II recommended dose (RP2D) | 27 weeks
  To evaluate the safety and tolerability of CYH33 and determine the maximum tolerated dose (MTD) and/or phase II recommended dose (RP2D) of CYH33 in adult and adolescent patients
Phase II PROS Cohort: BIRC-assessed objective response rate (ORR) at Week 24 | Baseline to 24weeks
  Proportion of patients achieving ≥20% reduction from baseline in the sum of target lesion volumes, with no progression of non-target lesions and no new lesions, as assessed by blinded independent review committee (BIRC).
Phase II PRVM Cohort: BIRC-assessed objective response rate (ORR) at Week 24 | Baseline to 24weeks
  Proportion of patients achieving ≥20% reduction from baseline in the sum of target lesion volumes, with no progression of non-target lesions and no new lesions, as assessed by blinded independent review committee (BIRC).

SECONDARY OUTCOMES:
Phase I: Pharmacokinetics of CYH33 and its metabolite I27 in the study population: Area Under the Curve from 0 to 24 hours (AUC0-24h) | Pre-dose and at 1, 2, 4, 6, 8, and 24 hours post-dose on Day 1 and Day 29.
  AUC0-24h of CYH33 and its metabolite I27 following drug administration will be assessed.
Phase I: Pharmacokinetics of CYH33 and its metabolite I27 in the study population: Maximum Concentration (Cmax) | Pre-dose and at 1, 2, 4, 6, 8, and 24 hours post-dose on Day 1 and Day 29.
  Cmax of CYH33 and its metabolite I27 following drug administration will be assessed.
Phase I: Pharmacokinetics of CYH33 and its metabolite I27 in the study population: Minimum Concentration (Cmin) | Pre-dose on Day 29.
  Cmin of CYH33 and its metabolite I27 following drug administration will be assessed.
Phase I: Pharmacokinetics of CYH33 and its metabolites in the study population: Time to Maximum Concentration (Tmax) | Pre-dose and at 1, 2, 4, 6, 8, and 24 hours post-dose on Day 1 and Day 29.
  Tmax of CYH33 and its metabolite I27 following drug administration will be assessed.
Phase I: Pharmacokinetics of CYH33 in the study population: Steady-State Apparent Clearance (CLss/F) | Pre-dose and at 1, 2, 4, 6, 8, and 24 hours post-dose on Day 1 and Day 29.
  CLss/F of CYH33 following drug administration will be assessed.
Phase I: The response rate and target lesion volume reduction rate as assessed by the investigators at each dose level | week 27
  A responder is defined as a ≥ 20% reduction in target lesion volume from baseline and in absence of progression of non-target lesions and without new lesions. The proportion of patients with reduced target lesion volume compared to baseline will also be assessed.
Phase I: The changes from baseline in the Brief Pain Inventory (BPI) Worst Pain Intensity Numerical Rating score at each dose level, based on the patient-reported outcome (PRO) diary | Up to approximately 48 months
  Pain is categorized into 11 levels from 0 to 10, where 0 indicates no pain at all and 10 indicates the most severe pain imaginable. Patients should assess and record their pain levels over the past 24 hours in the patient diary at each scheduled assessment visit.
Phase I: The changes from baseline in the Patient Global Impression of Change scale at each dose level, based on the patient-reported outcome (PRO) diary | Up to approximately 48 months
  Patients will compare their global impression of symptom changes with the pretreatment status, then categorize them into the following 7 grades: significantly relieved, moderately relieved, minimally relieved, no change, minimally worse, moderately worse, or significantly worse at each scheduled assessment visit.
Phase I: The changes from baseline in the quality of life scores at each dose level, based on the patient-reported outcome (PRO) diary | Up to approximately 48 months
  The Quality of Life Scale (EQ-5D-5L) consists of two parts. Part 1 assesses five quality-of-life-related indicators, with each indicator graded into five distinct levels for self-evaluation by the patient. Part 2 consists of patients' self-assessment of health status, with a maximum score of 100 points and a minimum score of 0 points.
Phase I: Frequency and severity of adverse events | Up to approximately 48 months
  The type, incidence, and severity of adverse events (AEs) (assessed according to the CTCAE Version 5.0 criteria).
Phase II : BIRC-assessed ORR at Week 48 (PROS cohort and PRVM cohort) | Week 48
  BIRC-assessed ORR at Week 48 (PROS cohort and PRVM cohort) Time Frame: From start of CYH33 treatment to Week 48
Phase II: BIRC-assessed ORR at Week 8 (Double-blind Period in PRVM cohort) | Week27
  BIRC-assessed ORR at Week 8 (Double-blind Period in PRVM cohort) Time Frame: From randomization to Week 8
Phase II: BIRC-assessed ORR at Weeks 8 and 16 (PROS cohort and PRVM cohort) | Weeks 8 and Week 16
  BIRC-assessed ORR at Weeks 8 and 16 (PROS cohort and PRVM cohort) Time Frame: From start of CYH33 treatment to Weeks 8 and 16
Phase II : Change from Baseline in Target Lesion Volume (PROS cohort and PRVM cohort) | Up to approximately 48 months
  Change from Baseline in Target Lesion Volume (PROS cohort and PRVM cohort) Time Frame: From start of CYH33 treatment to Week 48
Phase II: Investigator-assessed overall clinical response (PROS cohort and PRVM cohort) | Up to approximately 48 months
  Investigator-assessed overall clinical response (PROS cohort and PRVM cohort) Time Frame: From start of CYH33 treatment to Week 48
Phase II: Change from Baseline in Patient-Reported Outcomes (PROS cohort and PRVM cohort) | Up to approximately 48 months
  Change from Baseline in Patient-Reported Outcomes (PROS cohort and PRVM cohort) Time Frame: Up to approximately 48 months
Phase II: Safety and Tolerability of CYH33 (PROS cohort and PRVM cohort) | Up to approximately 48 months
  Safety and Tolerability of CYH33 (PROS cohort and PRVM cohort) Time Frame: Up to approximately 48 months
Phase II :Plasma Drug Concentrations of CYH33 and Metabolite I27 | Up to 5 cycles (approximately 20 weeks)
  Plasma Drug Concentrations of CYH33 and Metabolite I27

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Plastic Surgery Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Shanghai Ninth People Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan